CLINICAL TRIAL: NCT04039100
Title: Family Caregiver Ambassador Support for Family Caregivers of Patients With Hematological Disease (FAM CARE) - a Feasibility Study
Brief Title: Family Caregiver Ambassador Support for Family Caregivers of Patients With Hematological Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Iben Husted Nielsen, Principal Investigator, Ph.D.student, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: FAM CARE
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Multiple Myeloma; Lymphoma; Bone Marrow Transplantation; Neoplasms; Hematologic Diseases; Leukemia, Myeloid
Keywords: Peer to Peer; Psychosocial Support; Caregivers
MeSH Terms: conditions — Multiple Myeloma; Lymphoma; Neoplasms; Hematologic Diseases; Leukemia, Myeloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Family Caregiver Ambassador Support (Experimental): Intervention group: caregivers of newly diagnosed patients (n=30), former family caregivers as ambassadors (n=20)
  Interventions: Other: Family Caregiver Ambassador Support

INTERVENTIONS:
Other: Family Caregiver Ambassador Support — Family Caregiver Ambassador Support, with former caregivers of patients treated for hematological malignancies, being ambassadors for caregivers of newly diagnosed patients for a period of 12 weeks

SUMMARY:
Background: Family caregivers are of great importance to patients undergoing treatment for cancer, but at the same time, caregivers themselves are in great risk of distress and high symptom burden which affects their quality of life and ability to support the patients. Within hematology the context of treatment from hospital to home has changed in the past years placing more responsibilities on caregivers. Finding new ways to support caregivers within the health care context is important. Psychosocial interventions can enhance emotional well-being, and peer to peer support model has been found to be effective for patients coping with cancer. There is a lack of knowledge and evidence of the feasibility and effects of a peer-to-peer support in caregivers within hematology.

Aims: The study aim to examine the feasibility and safety of Family Caregiver Ambassador Support in caregivers of newly diagnosed patients with hematological disease, and to examine if it has an effects on symptoms and psychological wellbeing in both family caregivers and ambassadors. It is hypothesized that the family caregiver peer to peer support model will reduce symptoms of burden, reduce concerns and improve emotional and social well-being in family caregivers.

Design and methods: The study is a one arm feasibility intervention trial with family caregivers (n=30) and family caregiver ambassadors (N=20). Family Caregivers will be recruited at the Department of Hematology, Rigshospitalet. Family Caregivers will be partnered with a family caregiver ambassador. The intervention will be carried out in a 12-week period and consist of telephone and/or e-mail contact and face to face meetings with one follow-up at three months. Both caregiver and ambassador data will be collected at baseline, post intervention and follow-up 3 months.

Implication: The study has the potential to be a new model of care incorporated in the clinical setting to strengthen the support system for caregivers and may likely be tailored to other cancer groups and caregivers.

DETAILED DESCRIPTION:
Aim: To investigate whether a Family Caregiver Support Model intervention (FAM-CARE) is feasible and safe, and the impact on the caregiving role and psychosocial wellbeing in family caregivers of newly diagnosed patients with hematological malignancies, and former caregivers (family caregiver ambassadors).

Design and Methods: This study is a one arm feasibility 12-week intervention trial including family caregivers (FC) (n=30) and family caregiver ambassadors (FCA)(n=20).

Recruitment: FC will be recruited at the Department of Hematology, Rigshospitalet (RH). Eligible family caregivers will receive oral and written information on the project from main investigator Iben Husted Nielsen (IHN) within four weeks from the patients' diagnosis. Due to ethical considerations and data protection guidelines patients of eligible caregivers will be approached by IHN with permission to contact their caregivers before approaching them. Family caregivers will be given information on the study and the opportunity to raise questions and concerns and time to consider before enrollment.

FCA will be recruited voluntarily from the Department of Hematology, RH and patient associations (LyLe, Myeloma). The FCA is screened by IHN to assess their appropriateness for the intervention with interview questions regarding their motivation, availability, and vulnerability. They will be asked to sign a confidentiality commitment. The FCA will be informed that they must provide transportation but will receive a monetary incentive for their participation. Further FCA will be asked to provide information regarding age, gender, interests, work, education and social conditions and family role in order to match with the FC. FC and FCA will be matched according to their preferences i.e. patient diagnosis, age, gender and other factors that might create a mutual understanding and ease communication. Given the preferences cannot be granted, the FC and FCA will be involved in the decision.

FAM CARE Intervention: The intervention consists of individual support provided by the FCA to the FC, with minimum four face-to-face meetings between the FC and FCA, and with ad hoc telephone and/or email contact based on the FC's individual needs, and one follow-up telephone contact at 3 months. The place of meeting and purpose of each face-to-face meeting is agreed upon by the FC and FCA. The FCA will follow one FC at a time, however at the end of the 12- week period the FCA can choose to follow a new FC. Upon the first meeting and expectation agreement will be discussed between the FC and FCA. During the intervention the FCA will document the frequency of meetings, duration, place, content and quality of the interactions between FC and FCA.

Recruited FCA's will receive a six-hour group education and training program prior to interacting with FC. The training program include important and relevant actions and information on the role as ambassador, communication skills with emphasis on active listening, and discussion about volunteering and how to maintain appropriate boundaries to ensure that FCA are aware of their role as listeners who share their experiences only when solicited by the FC. The training will be organized by IHN and a project nurse and carried out by IHN, the project nurse and a project psychologist. To secure the safety of FCA during the intervention they will be offered to attend support meetings organized by IHN and the project psychologist to process and share their experiences with being an ambassador. Support meetings will be held every second month and FCA can request individual supervision from the project psychologist during the intervention. Any severe adverse events will be documented and acted upon.

Outcome measures and data collection: Data are collected by patient reported outcome measures (PROM) as self-reported questionnaires completed by FC electronically prior to intervention, post intervention (12-weeks) and at 3-month follow-up. PROM is completed by FCA prior to intervention and at post intervention (12 weeks). Socio-demographic data are collected by questionnaire. At the end of the 3-months follow-up focus group interviews with FC and FCA will be conducted on their experiences.

ELIGIBILITY:
Inclusion Criteria:

* Eligible family caregivers (FC) are ≥ 18 years old and a family member or significant other of a patient with hematological malignancy in one of three categories: 1) acute: newly diagnosed with acute leukemia/high risk myelodysplastic syndrome (MDS) or lymphoma ≤ 4 weeks from diagnosis who will receive intensive chemotherapy (n=10), 2) chronic: diagnosed with myeloma or chronic leukemia/MDS or lymphoma to receive less intensive chemotherapy or palliation (n=10) and 3) complex course of treatment: to undergo a stem cell transplantation (n=10).
* Eligible Family Caregiver Ambassadors (FCA) are ≥18 years old and a family caregiver of a survivor of a patient with hematological malignancy (in complete remission) and provides consent to participate in the ambassador training program. Informed written consent will be provided by all participants

Exclusion Criteria:

* Participants (FC and FCA) will be excluded if they do not understand, read and speak Danish, if they have unstable medical disease or cognitive/psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Up to 2 years
  Number of participants included from eligible family caregivers
Adherence to intervention | up to 24 weeks
  Number of weeks completed out of planned weeks of intervention
Emotional reactions (quality of contacts) | up to 24 weeks
  Registration on descriptive data on content of contacts with project team members (primary investigator/project psychologist/project nurse)
Emotional reactions (numbers of contacts) | up to 24 weeks
  Registration on numbers of contacts with project team members (primary investigator/project psychologist/project nurse)

SECONDARY OUTCOMES:
Depression | Change measures (baseline, 12 weeks, 24 weeks)
  Measured with the Hospital Anxiety and Depression Scale (HADS)
Anxiety | Change measures (baseline, 12 weeks, 24 weeks)
  Measured with the Hospital Anxiety and Depression Scale (HADS)
Sleep | Change measures (baseline, 12 weeks, 24 weeks)
  Measured with the Pittsburgh Sleep Quality Index (PSQI)
Health-related quality of life | Change measures (baseline, 12 weeks, 24 weeks)
  Measured with the Short form-36 (SF-36)
Self-efficacy | Change measures (baseline, 12 weeks, 24 weeks)
  Measured with the General Self-Efficacy Scale questionnaire. Scale ranges with total scores (higher scores indicating better self-efficacy)
Caregiver roles and responsibilities | Change measures (baseline, 12 weeks, 24 weeks)
  Measured with the Caregiver Roles and Responsibilities Scale (CRRS) questionnaire measuring cancer impact on the lives of caregivers, each subscale provided by total scores
Number of contacts between family caregiver and ambassador | Up to 12 weeks
  Measured by the total number of contacts during the planned weeks of intervention.
Length of contacts between family caregiver and ambassador | Up to 12 weeks
  Measured by the total time of contacts during the planned weeks of
Thematic content of the contacts between family caregiver and ambassador | Up to 12 weeks
  Measured by ambassadors registrations and descriptions of thematic content of the contacts with the family caregiver

CONTACTS AND LOCATIONS:
Overall Officials: Mary Jarden, ph.d., Study Director — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Østerbro, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Noerskov KH, Nielsen IH, Rahbaek ES, Halbro S, Mortensen AO, Overgaard UM, Piil K, Jarden M. Implementation and Evaluation of Peer Ambassador Support to Patients Newly Diagnosed With Hematological Cancer and Their Caregivers. Nurs Res Pract. 2025 Apr 28;2025:4528051. doi: 10.1155/nrp/4528051. eCollection 2025. PMID 40330711
- [Derived] Husted Nielsen I, Piil K, Tolver A, Gronbaek K, Kjeldsen L, Jarden M. Family caregiver ambassador support for caregivers of patients with newly diagnosed hematological cancer: a feasibility study. Support Care Cancer. 2022 Aug;30(8):6923-6935. doi: 10.1007/s00520-022-07089-0. Epub 2022 May 11. PMID 35543814